CLINICAL TRIAL: NCT01664013
Title: The Impact of Botulinum Toxin Treatment in Quality of Life of Cervical Dystonia Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Roongroj Bhidayasiri (Other)
Responsible Party: Sponsor-Investigator, Roongroj Bhidayasiri, Associate Professor, Chulalongkorn University
Organization: Chulalongkorn University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT_IT_010
Record Dates: First submitted 2012-08-07; First posted 2012-08-14 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Botulinum Toxin; Quality of Life; Cervical Dystonia
MeSH Terms: conditions — Torticollis | interventions — Botulinum Toxins, Type A

ARMS (1):
- Neuronox (Experimental): Neuronox® is a botulinum toxin type A (BoNT/A) product developed by Medytox Inc. (Medytox) of Korea. Neuronox® was first approved by the Korean Food and Drug Administration in 2006, and by Thai Food and Drug Administration in 2008.
  Interventions: Drug: Nuronox

INTERVENTIONS:
Drug: Nuronox — Reconstituted Neuronox® is injected at a dose determined by the physician based upon his/her clinical experience with botulinum toxin.Actual dose and injection site should be adjusted individually considering the muscle mass, degree of spasticity, body weight, and response to any previous botulinum toxin injections.
  Other Names: Clostridium Botulinum Toxin A

SUMMARY:
The purpose of this study is to investigate the impact of botulinum toxin treatment in quality of life(QoL) in cervical dystonia patients

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 18 years to 75 years
* Subjects requiring treatment for a clinical diagnosis of cervical dystonia
* Willing to provide written informed consent before any study-related procedures.

Exclusion Criteria:

* Patients with pure anterocollis
* Patients with an anaphlyactic response history to botulinum toxin type A.
* Patients who have been treated with botulinum toxin type A within 3 month.
* Females who are pregnant, planning pregnancy, unable to use contraception or lactating.
* Any medical condition that may put the subject at increased risk with exposure to botulinum toxin at the discrimination of investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
To investigate the change of quality of life of cervical dystonia patients after botulinum toxin treatment measured by CDQ-24. | 6 weeks
  To investigate the change of quality of life of cervical dystonia patients from baseline at 6 weeks after botulinum toxin treatment measured by CDQ-24.

SECONDARY OUTCOMES:
To investigate the change of QoL of cervical dystonia patientsafter botulinum toxin treatment measured by SF-36 (Thai version) | 6 weeks
  To investigate the change of QoL of cervical dystonia patients at 6weeks after botulinum toxin treatment from baseline measured by SF-36 (Thai version).
To Investigate the change of symptom after botulinum toxin treatment measured by TWSTRS score | 6 weeks
  To Investigate the change of symptom at 6weeks after botulinum toxin treatment from baseline measured by TWSTRS score

CONTACTS AND LOCATIONS:
Locations (1):
- Roongroj Bhidayasiri, Pathumwan, Bangkok, Thailand